CLINICAL TRIAL: NCT06791967
Title: Effectiveness of a Home-base Walking Exercise Program on Depression,Frailty,and Quality of Life in Patients with Heart Failure: a Single-Center Randomized-Controlled Trial
Brief Title: The Impact of a Home-Based Walking Exercise Program on Heart Failure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202407218RIND
Record Dates: First submitted 2025-01-12; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-09

CONDITIONS: Heart Failure; Home-based Walking Excercise; Depression; Frailty; Quality of Life
MeSH Terms: conditions — Heart Failure; Depression; Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Home-based walking group (Experimental): In addition to general health education, patients will receive a 12-week home walking exercise program intervention after discharge.
  Interventions: Behavioral: home-based walking program
- General health education group (No Intervention): A general routine health education in the hospital before discharge.

INTERVENTIONS:
Behavioral: home-based walking program — The home-based walking intervention involves five walking sessions per week over 12 weeks, with a target of 3,000 additional steps per session beyond daily activities. In the first week, participants in the experimental group will wear a smart wristband upon waking to record their average daily steps, which will guide their walking goals. By the 7th week, participants are expected to achieve at least 3,000 extra steps per session, completed in 30 continuous minutes. The wristband, synced via Bluetooth to its companion app, can store up to one month of walking data. Weekly phone follow-ups will record participants' daily step counts. No additional cloud uploads of personal data are required.
  Arms: Home-based walking group

SUMMARY:
Heart disease is the second leading cause of death in Taiwan, with approximately 700,000 individuals affected by heart failure. Despite the proven benefits of rehabilitative exercise, participation in cardiac rehabilitation remains suboptimal. To address this, integrating physical activity into daily life, such as home-based walking exercises, offers a practical alternative to promote health and improve outcomes in heart failure patients. Walking exercises have been shown to significantly impact mortality rates and enhance the quality of life in this population.

This study aims to assess the effects of a 12-week home-based walking exercise program on depression, frailty, and quality of life in patients with heart failure. Using an experimental design, heart failure patients hospitalized in a medical center's internal medicine ward were randomly divided into an experimental group (n=34) and a control group (n=34). While both groups received standard health education, the experimental group also participated in a home-based walking intervention after discharge. Data were collected before the intervention and at the 1st and 3rd months post-intervention. The generalized estimation equation (GEE) was employed to analyze changes in depression, frailty, and quality of life, focusing on group differences and interactions between time and group.

The expected outcomes of the study include improved quality of life, reduced frailty, and alleviated depression in the experimental group, highlighting the value of home-based walking exercise. Additionally, the intervention model can complement existing post-discharge nursing practices by incorporating remote nursing guidance to enhance exercise adherence without increasing healthcare costs. This approach not only benefits patients by encouraging long-term physical activity but also reduces the burden on healthcare systems, making it a sustainable and effective strategy for managing heart failure.

DETAILED DESCRIPTION:
Background: According to statistics from the Ministry of Health and Welfare, heart disease ranks second among the top ten causes of death in the nation. It is estimated that approximately 700,000 people in Taiwan suffer from heart failure. Despite research confirming the multiple benefits of rehabilitative exercise, actual patient participation in rehabilitation is not ideal. Therefore, incorporating physical activities from daily life as an alternative method can promote the clinical value and practical significance of home-based walking exercise. Walking exercise has a significant impact on the mortality rate and quality of life of patients with heart failure.

Objective: This study aims to investigate the benefits of a home-based walking exercise intervention on depression, frailty, and quality of life in patients with heart failure.

Methods: The study adopts an experimental research design, targeting heart failure patients hospitalized in the internal medicine ward of a medical center in northern Taiwan. Participants were randomly assigned to either the control group (n=34) or the experimental group (n=34). In addition to receiving standard health education, the experimental group participated in a 12-week home-based walking exercise program after discharge. The control group received standard health education once before discharge. Data were analyzed using the generalized estimation equation (GEE) to examine the variables of depression, frailty, and quality of life in both the experimental and control groups before the intervention, and at the 1st and 3rd months post- intervention. The analysis focused on group effects and the interaction between group and time.

Expected Clinical Practice Applications: Based on past literature analysis, home-based walking exercise combined with remote nursing guidance is expected to improve the quality of life, reduce frailty, and alleviate depression in patients with heart failure. Patients can significantly benefit from performing walking exercises at home, while also reducing the clinical workload and costs associated with cardiac rehabilitation for healthcare providers. The intervention model from this study can coexist with current post-discharge nursing follow-up practices. By encouraging continuous home-based walking exercises through remote nursing guidance, the approach ensures ongoing care and personalized nursing without incurring additional nursing costs, thereby effectively enhancing patients' willingness to engage in exercise.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with heart failure classified as New York Heart Association (NYHA) Functional Class II-III by a physician.
* Approval from the attending physician to participate in the home-based walking program after discharge.
* Aged between 18 and 80 years.
* Patients unable to attend outpatient cardiac rehabilitation.
* No regular exercise habits, such as performing less than 30 minutes of aerobic exercise per week.
* Able to walk independently without the aid of assistive devices.
* Patients with clear consciousness, no cognitive impairment, and no history of mental illness.
* Able to communicate in Mandarin or Taiwanese dialect.
* Willing to participate in the study, sign the informed consent form, and comply with the home-based walking program.

Exclusion Criteria:

* Patients diagnosed with heart failure classified as New York Heart Association (NYHA) functional class IV by a physician.
* Patients diagnosed with depression by a psychiatrist.
* Patients with cognitive impairment or language communication disorders.
* Patients who are bedridden for an extended period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Depression (Patient Health Questionnaire-9,PHQ-9) | baseline, 1 month, 3 months
  A state of mood in daily life characterized by a loss of interest or pleasure in activities, accompanied by symptoms such as weight loss or decreased appetite, insomnia or excessive sleep, psychomotor abnormalities or agitation, fatigue or lack of energy, excessive guilt or self-deprecation, difficulty concentrating or making decisions, and suicidal thoughts, plans, or behaviors.
  Scoring Method： Each response is assigned a score based on the following scale:0 points: Not at all,1 point: Several days,2 points: More than half the days,3 points: Nearly every.
  PHQ-9 score obtained by adding score for each question (total points). 0-4: Minimal or no depression 5-9: Mild depression 10-14: Moderate depression 15-19: Moderately severe depression 20-27: Severe depression Higher scores indicate more severe depressive symptoms, with a score of 10 or above generally suggesting the need for further clinical evaluation or intervention.
Frailty (CSHA-CFS) | baseline, 1 month, 3 months
  Frailty is defined as a decline in overall physiological resilience, making it difficult to cope with stress or even daily activities. The current criteria for identifying frailty include the presence of at least three of the following five symptoms: reduced grip strength, decreased energy levels, slow walking speed, insufficient physical activity.
  A score from 1 (very fit) to 9 (terminally ill) is given based on the descriptions and pictographs of activity and functional status.
  Scoring Description:
  1. Very Fit
  2. Fit
  3. Managing Well
  4. Living with Very Mild Frailty
  5. Living with Mild Frailty
  6. Living with Moderate Frailty
  7. Living with Severe Frailty
  8. Living with Very Severe Frailty
  9. Terminally Ill In the CSHA-CFS assessment, higher scores indicate greater frailty. A score of 1 reflects very fit individuals, while a score of 9 indicates terminal illness and full dependency. Mid-range scores (4-6) signify moderate frailty with functional limitations.
Quality of Life (Minnesota Living With Heart Failure Questionnaire,MLHFQ) | baseline, 1 month, 3 months
  Quality of life refers to an individual's functional abilities and well-being across physical, psychological, and social domains. Functionality includes physical functions such as self-care (e.g., bathing, dressing, walking); role functions, such as work-related activities like household chores and professional tasks; and social functions, which involve the extent of interaction with family and friends. Well-being, on the other hand, is more subjective than functionality and encompasses emotions such as happiness, sadness, depression, anxiety, pain, and fatigue.
  Scoring Range: The MLHFQ consists of 21 items, each scored on a scale from 0 to 5.
  0: No impact on daily life. 5: Maximum impact on daily life. Total Score: Add the scores for all 21 items to calculate the total score. The total score ranges from 0 to 105, with higher scores indicating a greater negative impact of heart failure on the patient's quality of life.

IPD SHARING:
Plan to Share IPD: No